CLINICAL TRIAL: NCT06814821
Title: Web-based Rehabilitation After Surgical Salvage Procedures for Wrist Osteoarthritis: a Randomized Controlled Trial
Brief Title: Web-based Rehabilitation After Surgical Salvage Procedures for Wrist Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Elin Swärd, Principal Investigator, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Web-based rehab - wrist OA
Record Dates: First submitted 2024-11-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Wrist Osteoarthritis
Keywords: web-based rehabilitation; wrist osteoarthritis; SLAC; SNAC; exercise therapy; arthritis; randomized controlled trial
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-based rehabilitation (Experimental): The web-based platform contains text, images, and videos which will educate and inform the patient regarding the operation and rehabilitation.
  There will be no scheduled physical consultations, however participants may request additional video consultations and can send text messages to the hand therapist.
  Interventions: Other: Web-based rehabilitation
- Standard rehabilitation (Active Comparator): The control group receive the same education and exercises. The information is provided verbally and a booklet with images of the exercises is given. However, they do not get access to the web-based platform and follow-up appointments are face-to-face at the clinic.
  At the follow-up appointments, participants perform their exercises, and adjustments and corrections are made when needed.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Web-based rehabilitation — Participants perform their rehabilitation independently with the instructions from the web-based platform.
  Arms: Web-based rehabilitation
Other: Standard rehabilitation — Participants attend physical visits at the clinic to get instructions and support in their rehabilitation. Written and verbal instructions will be given.
  Arms: Standard rehabilitation

SUMMARY:
Wrist osteoarthritis is often caused by past trauma to the wrist. The primary symptom is joint pain. Salvage surgery is the final solution if exercise therapy, analgesics, orthoses, or cortisone injections fail to relieve pain.

This trial aims to evaluate if a web-based rehabilitation protocol is non-inferior to standard, face-to-face, rehabilitation in terms of patient-reported outcome after surgical salvage procedures.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic disease which affects all tissues of the joint - cartilage, ligaments, synovial membrane, tendons, and bone. The primary symptom is joint pain but other symptoms like swelling, stiffness, crepitus, and joint instability may also be present.

OA is most in common in knee, hip, and hand but all joints can be affected. It is estimated that nearly 50% of women and 25% of men risk hand OA during their lifetime. Interphalangeal joints and thumb base are the primarily affected joints in the hand while the wrist is less common. Wrist OA is, in contrary to interphalangeal joints and thumb base, more common in men than in women and at a younger age.

Wrist OA is often caused by past trauma to the wrist e.g., fractures, dislocations, and ligament injuries. However, avascular necrosis i.e., Mb Kienböck and Mb Preiser, and other medical conditions may also lead to wrist OA.

Although there is no cure, patients with hip and knee OA, may benefit from self-management treatment options. For hand and wrist OA, the effects of exercise therapy are less studied. A Cochrane review found low-quality evidence of small positive effects of exercise on pain, function, and finger joint stiffness. In wrist OA, a recent randomized controlled trial reported that neuromuscular joint-protective exercise therapy was not superior to range of motion exercises in reducing pain and improving function.

Salvage surgery is the final solution if exercise therapy, analgesics, orthoses, or cortisone injections fail to relieve pain. Numerous studies describe different types of surgical salvage procedures in wrist OA but, to our knowledge, none compare different types of rehabilitation after surgery.

Telerehabilitation for acute and chronic musculoskeletal disorders including OA have been used for over a decade, with an increased demand during the Covid 19 pandemic, and continue to evolve. Telerehabilitation is defined as the "Delivery of therapeutic rehabilitation at a distance or offsite using telecommunication technologies" and includes a wide variety of interventions such as assessments, education, or exercises via mobile or tablet applications, web pages and so forth.

Systematic reviews have shown telerehabilitation to be equal to or superior to standard rehabilitation in various musculoskeletal conditions but without a high level of evidence. Few previous studies focus on disorders of the hand and wrist. In conservatively treated hand OA, operated carpal tunnel syndrome, and operatively and nonoperatively treated patients with bony or soft tissue conditions of the hand and wrist, mobile applications were better than home exercise programs on paper in improving upper limb function and decreasing the number of clinical appointments and referral for rehabilitation.

Telerehabilitation after OA surgery has shown good results in both patient satisfaction and clinical outcomes, but previous studies have mainly focused on hip and knee OA. Although a steadily increasing number of studies, investigators have not been able to find any studies comparing web-based or telerehabilitation to standard, face-to-face, rehabilitation after surgical salvage procedures for wrist OA.

Research question:

Is a web-based rehabilitation protocol non-inferior to standard, face-to-face, rehabilitation in terms of patient-reported outcome after surgical salvage procedures for wrist osteoarthritis?

Hypothesis:

A postoperative web-based rehabilitation protocol is non-inferior to standard rehabilitation in terms of patient-reported outcome measured by Patient Reported Wrist Evaluation (PRWE) 3 months after cast removal in patients operated with surgical salvage procedures for wrist osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery:
* Four corner fusion (4CF)
* Lunate-Capitate fusion (LCF)
* Scaphoid-Trapezium-Trapezoid fusion (STT)
* Radius-Scaphoid-Lunate fusion (RSL)
* Proximal Row Carpectomy (PRC)
* Access to digital identification.

Exclusion Criteria:

* Unstable rheumatoid arthritis or other chronic inflammatory arthritis. However, stable inflammatory arthritis with unchanged medication during the last 12 weeks is not an exclusion criteria.
* History of psoriasis arthritis, gout, or pseudogout affecting the hand or wrist.
* Symptomatic OA in nearby joints.
* Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction, inability to use web-based tools).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) score, 3 months after cast removal compared to baseline. | From enrollment to the end of treatment at 3 months after cast removal.
  Patient Rated Wrist Evaluation (PRWE) score (0-100 points). A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Pain at rest and on load - change in score from baseline to cast removal and 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  Pain Numerical Rating Scale (PNRS). A higher score indicates a worse outcome.
Quality of life (EQ-5D-5L) - change in score from baseline to cast removal and 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  EQ-5D-5L (0-1 points). A lower score indicates a worse outcome.
Pain catastrophizing scale - change in score from baseline to cast removal and 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  Pain catastrophizing scale (PCS) (0-52 points). A higher score indicates a worse outcome.
Tampa Scale of Kinesiophobia - change in score from baseline to cast removal and 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  Tampa Scale of Kinesiophobia (TSK-17) (17-68 points). A higher score indicates a worse outcome.
Range of motion - change from baseline to cast removal and 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  Range of motion (ROM) of the wrist (extension/flexion, radial/ulnar deviation, pronation/supination).
Grip strength - change in score from baseline to 3 months after cast removal. | From enrollment to the end of treatment at 3 months after cast removal.
  Grip strength (hydraulic hand dynamometer)
Patient Reported Experience Measures (PREM). | 3 months after cast removal.
  * Are you satisfied with how you can contact your healthcare provider?
  * Did you receive enough information about your surgery and rehabilitation?
  * Do you feel that your rehabilitation needs have been met?
  * Are you satisfied with your rehabilitation?
Adherence to excercise program. | From enrollment to the end of treatment at 3 months after cast removal.
  Adherence, using an exercise diary.
Complications - number of participants. | From enrollment to the end of treatment at 3 months after cast removal.
  E.g complex regional pain syndrome,
Length of sick leave, ability to return to previous work. | From enrollment to the end of treatment at 3 months after cast removal.
Number of consultations. | From enrollment to the end of treatment at 3 months after cast removal.
  Number of face-to-face consultations in standard rehabilitation group. Number of face-to-face and video consultations in web-based group.
Differences in direct costs - between groups. | From enrollment to the end of treatment at 3 months after cast removal.
  Differences in direct costs associated with treatment and indirect costs e.g., sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Elin M Swärd, PhD, Principal Investigator — KI Department of Clinical Science and Education, Södersjukhuset

IPD SHARING:
Plan to Share IPD: No